CLINICAL TRIAL: NCT04123119
Title: Development of a Live Attenuated Rotavirus Vaccine as a Human Infection
Brief Title: Development of a Live Attenuated Rotavirus Vaccine as a Human Infection Challenge Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Imperial College London (Other); Christian Medical College, Vellore, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HicVac Rota
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Diarrhoeal Disease
MeSH Terms: interventions — Rotavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rotarix Arm (Experimental)
  Interventions: Biological: Rotavirus vaccine

INTERVENTIONS:
Biological: Rotavirus vaccine — An exploratory and observational cohort study following infants receiving two standard doses of live, attenuated, oral Rotarix™ administered at 6 & 10 weeks.

SUMMARY:
The impact of licensed rotavirus vaccines in LMICs is limited by their lower immunogenicity and efficacy in these settings. Improved vaccines and vaccination schedules would result in substantially greater reductions in infant diarrhoeal disease and mortality. Placebo-controlled trials of new rotavirus vaccines are no longer ethical, leading to challenges for traditional routes of licensure for vaccines that are in the development pipeline.

A HIC model of rotavirus would address these challenges, whilst also offering an opportunity to study the causes of poor oral vaccine immunogenicity. Rotarix™ is in routine use in Zambia administered at 6 and 10 weeks infant age. Shedding of rotavirus vaccine after vaccination has recently been explored as a measure of mucosal immunity, analogous to oral poliovirus vaccine challenge models.

We propose to explore methodological development of an attenuated vaccine as a HIC model to advance rotavirus immunology and vaccinology in Zambian infants. We will evaluate use of minimally invasive procedures including sublingual/submandibular sampling and stool collection for viral shedding as measures of vaccine-induced and naturally acquired mucosal immunity. This approach holds the potential to develop the first rotavirus HIC model in a low-income country and could be used to accelerate licensure of new rotavirus vaccines and explore causes of poor oral vaccine efficacy as well as correlates of vaccine protection.

To do this, we will recruit a cohort of 22 Zambian infants receiving Rotarix™ at 6 and 10 weeks as part of their routine immunisation. Infants will be followed up actively on the day of vaccination, days 1,3,5 and 7 following each vaccine dose for collection of stool and saliva samples. Blood samples for IgA and IgG titres will be collected on days 0, 28, 31 and 56, and standard ELISA methods used to determine vaccine seroconversion.

The work brings together collaborators at the Centre for Infectious Disease Research in Zambia, Imperial College in UK and Christian Medical College, Vellore in India to prepare the Zambian centre as a potential HIC model site.

DETAILED DESCRIPTION:
Diarrhoeal disease is a leading cause of morbidity and mortality in young children, particularly those living in the developing countries of South Asia and sub-Saharan Africa1. Rotavirus is the most common causative agent of moderate to severe diarrhoea in children under age five, responsible for an estimated 215,000 infant deaths every year, most of which occur within lower and middle-income countries (LMICs)2. The widespread introduction of two World Health Organisation (WHO)-approved rotavirus vaccines , RotarixTM, (GlaxoSmithKline Biologicals, Belgium) and RotaTeq, (Merck and Co, New Jersey), has contributed substantially to reducing the number of rotavirus-associated hospitalisations and deaths3-18. However, even with these gains, rotavirus vaccines have repeatedly demonstrated lower immunogenicity, effectiveness, efficacy and duration of protection in children living in LMICs as compared to high-income countries19,20,21. Thus, even after the introduction of rotavirus vaccines (RV), rotavirus remains the leading cause of diarrhoeal morbidity and mortality within these settings. Improved RV would result in substantially greater reductions in diarrhoeal disease morbidity and mortality among infants; there is, therefore, an urgent need to understand the reduced performance of currently available live attenuated oral vaccines in LMICs, to inform and accelerate the development of maximally effective therapeutics.

Recent studies have suggested that alternative schedules could also enhance immunogenicity and eventual vaccine performance in LMICs22,23. In addition, new RV candidates with alternative routes of administration are under development, and show promise for improved vaccine performance21,24,25. However, traditional pathways for licensure of new vaccines that are in the development pipeline through clinical trials have become challenging, with placebo-controlled trials no longer considered ethical, and field efficacy trials requiring increasingly larger cohorts to compare new candidates against existing vaccines. Human Infection Challenge (HIC) models have historically been employed to accelerate vaccine development and offer an opportunity to study both pathogenesis and vaccine immunogenicity mechanisms particularly in human-restricted pathogens. HIC models have not been widely used and accepted in LMICs even though there are scientific and ethical merits of considering the unique opportunity this methodology offers.

We propose to explore the methodological development of an attenuated vaccine as a HIC model to advance rotavirus immunology and vaccinology in Zambian infants. We will also evaluate the use of minimally invasive procedures, including collection of saliva for antibody measurement and stool samples for vaccine virus shedding as measures of vaccine-induced mucosal immunity.

Objective 1 To profile rotavirus specific IgA and IgG responses to vaccination and determine correlation between serum and saliva.

Specific Objective 1a: To profile rotavirus specific IgA and IgG responses at baseline (Day 0), pre-dose 2 (day 28) and 1 month post dose 2 (day 56) in serum and saliva to determine seropositivity and vaccine seroconversion.

Objective 2 To profile cytokine immune responses and determine correlation between serum and saliva.

Specific objective 2a: Determine cytokine profiles in serum and saliva at baseline (Day 0) and track their association with vaccine seroconversion (day 56).

Specific objective 2b: To profile cytokine responses immediately before dose 2 vaccination (day 28), and at 3 days after administration of the second vaccine dose (day 31: rotavirus vaccine challenge).

Objective 3: To assess the relationship of antibody levels in serum and saliva at the time of vaccination (day 0) and on days 28, 31, and 56, against faecal shedding of RV strain in stool collected and on days 3,5,7,14 and 21, and also on day 28 and post dose 2 vaccination days 31, 33, 35, 42, 49 and 56.

Objective 4: To profile and characterize the immediate cytokine immune response to the vaccine in saliva collected on day 0 and day 31, in order to determine whether saliva could serve as a satisfactory proxy for serum in evaluating vaccine-induced mucosal immunity.

1. Methodology

1. Study Design An exploratory and observational cohort study following infants receiving two standard doses of live, attenuated, oral Rotarix™ administered at 6 & 10 weeks. Infants will be enrolled during the routine EPI visit for week 6 immunizations following administration and provision of written informed consent by their mothers/legal guardians. Each infant will remain in the study for up to 56 days during which they will be intensively followed up with study activities and/or scheduled study clinic visits (summarized in Table 1 below).
2. Study site and population The study will be conducted at George Clinic in Lusaka where the government maternal child health (MCH) and antiretroviral therapy (ART) clinics as well as the CIDRZ George Clinical Study Site are co-located. George Clinic has a catchment population of 145,23053 and is located in a typical peri-urban setting in Lusaka within a surrounding slum. We plan to recruit participants as they randomly attend the health facility. CIDRZ has a good research facility already existing at this clinic and below is a schematic image of the site plan.
3. Selection of participants, sampling methods and sample size Sample size Considerations Participants will be randomly selected from mother-infant pairs attending routine antenatal care at George Clinic. As this will be an exploratory and methodological development study, no formal sample size calculations have been undertaken. We have pragmatically decided to enroll 20 infants which is generally acceptable for phase I-type studies. In case of an estimated 10% attrition due to loss to follow up, we have adjusted the sample to recruit 22 infants.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants as established by medical history and clinical examination before entering study
* age: > 6 and <8 weeks at the time of enrollment
* parental ability and willingness to provide informed consent
* parental intention to remain in the area with the child during the study period.

Exclusion Criteria:

* Presence of fever on the day of enrollment
* Acute disease at the time of enrollment
* Concurrent participation in another clinical trial throughout the entire timeframe for this study
* Presence of malnutrition or any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination that would compromise the participant's health or is likely to result in nonconformance to the protocol
* History of premature birth (<37 weeks gestation)
* History of congenital abdominal disorders, intussusception, or abdominal surgery
* Known or suspected impairment of immunological function based on medical history and physical examination
* Prior receipt of rotavirus vaccine
* A known sensitivity or allergy to any components of the study vaccine
* History of anaphylactic reaction
* Major congenital or genetic defect
* Participant's parents not able, available or willing to accept active follow-up by the study staff
* Has received any immunoglobulin therapy and/or blood products since birth or planned administration during the study period
* History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including corticosteroids.
* Any condition in the parents/infant that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parents' ability to give informed consent.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Measurement of serum RV-IgA and RV-IgG | 3 months
  Four (4) fold change in Serum anti-rotavirus specific IgA titles at 3 months post dose two

SECONDARY OUTCOMES:
Assessment of Viral shedding in stool | 5 months
  rotavirus NSP2 specific reverse transcription polymerase chain reaction (RT- PCR) in stool samples
Measurement of cytokines | 5 months
  cytokine profiling on serum and saliva

CONTACTS AND LOCATIONS:
Overall Officials: Roma Chilengi, MBCHB, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- George Clinical Research Site, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No